CLINICAL TRIAL: NCT00280566
Title: A Phase 3, Randomized, 6-Month, Double-Blind Trial in Subjects With Bipolar I Disorder to Evaluate the Continued Safety and Maintenance of Effect of Ziprasidone Plus a Mood Stabilizer (vs Placebo Plus a Mood Stabilizer) Following a Minimum of 2 Months of Response to Open-Label Treatment With Both Agents
Brief Title: Safety and Maintenance of Effect of Ziprasidone Plus a Mood Stabilizer in Bipolar I Disorder (Manic or Mixed)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A1281137
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Results first posted 2009-12-14 (Estimated); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Bipolar Mania; Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — ziprasidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ziprasidone (Experimental): Active treatment, double-blind, randomized arm
  Interventions: Drug: Ziprasidone Oral Capsule
- Placebo (Placebo Comparator): Placebo treatment, double-blind, randomized arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Oral capsule formulation: Patients will be treated initially with open-label ziprasidone in the range of 40-80 mg BID (twice a day) for at least 10 weeks and up to 16 weeks. Patients who achieve a stable treatment regimen and whose symptoms stabilize for 8 consecutive weeks by Week 16 (Week 10 at the earliest) will be randomized. Patients randomized to placebo will be tapered off the open-label ziprasidone by 20 mg BID every 2 days (in a double-blinded manner) until they are completely off ziprasidone and are on matching placebo capsules for up to 24 weeks of double-blind treatment.
  Arms: Placebo
Drug: Ziprasidone Oral Capsule — Oral capsule formulation: Patients will be treated initially with open-label ziprasidone in the range of 40-80 mg BID for at least 10 weeks and up to 16 weeks. Patients who achieve a stable treatment regimen and whose symptoms stabilize for 8 consecutive weeks by Week 16 (Week 10 at the earliest) will be randomized. Patients randomized to ziprasidone will continue to receive the same stable treatment regimen achieved during the open-label treatment, ie, either 40 mg BID, 60 mg BID or 80 mg BID for up to 24 weeks of double-blind treatment.
  Other Names: Geodon, Zeldox
  Arms: Ziprasidone

SUMMARY:
The purpose of this study is to determine if ziprasidone plus a mood stabilizer will continue to be a safe and effective treatment regimen for adults with Bipolar I Disorder (manic or mixed symptoms) after they have achieved 8 consecutive weeks of symptom improvement on the regimen.

ELIGIBILITY:
Inclusion Criteria:

Adults meeting DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition) criteria for Bipolar I Disorder (currently with manic or mixed symptoms)

Exclusion Criteria:

Ultra rapid cyclers and subjects with significant cardiovascular disease including history of QT prolongation and/or congenital long QT syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2005-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (92):
- United States (62):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Costa Mesa, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, National City, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Temecula, California
  - Pfizer Investigational Site, Altamonte Springs, Florida
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Maitland, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, North Miami, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Tavares, Florida
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Smyrna, Georgia
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Des Plaines, Illinois
  - Pfizer Investigational Site, Libertyville, Illinois
  - Pfizer Investigational Site, Naperville, Illinois
  - Pfizer Investigational Site, Oak Brook, Illinois
  - Pfizer Investigational Site, Schaumburg, Illinois
  - Pfizer Investigational Site, Terre Haute, Indiana
  - Pfizer Investigational Site, Topeka, Kansas
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Owensboro, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Rockville, Maryland
  - Pfizer Investigational Site, Pittsfield, Massachusetts
  - Pfizer Investigational Site, Taunton, Massachusetts
  - Pfizer Investigational Site, Olive Branch, Mississippi
  - Pfizer Investigational Site, Ridgeland, Mississippi
  - Pfizer Investigational Site, Saint Charles, Missouri
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Nashua, New Hampshire
  - Pfizer Investigational Site, Paramus, New Jersey
  - Pfizer Investigational Site, Teaneck, New Jersey
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Olean, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Bethany, Oklahoma
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Media, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Arlington, Texas
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Bellaire, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, DeSoto, Texas
  - Pfizer Investigational Site, Houston, Texas
- Chile (2):
  - Pfizer Investigational Site, Santiago, RM
  - Pfizer Investigational Site, Santiago
- France (4):
  - Pfizer Investigational Site, Angoulême
  - Pfizer Investigational Site, Brest Naval
  - Pfizer Investigational Site, Douai
  - Pfizer Investigational Site, Mulhouse
- Germany (3):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Cham
  - Pfizer Investigational Site, Essen
- Pfizer Investigational Site, Guatemala City, Guatemala
- Pfizer Investigational Site, New Territories, Hong Kong
- India (7):
  - Pfizer Investigational Site, Ellisbridge, Ahmedabad
  - Pfizer Investigational Site, Tirupati, Andhra Pradesh
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Mysore, Karnataka
  - Pfizer Investigational Site, Chennai, Tamil Nadu
  - Pfizer Investigational Site, Ludhiana
  - Pfizer Investigational Site, Pune
- Italy (4):
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Parma
  - Pfizer Investigational Site, Pisa
- Mexico (2):
  - Pfizer Investigational Site, Zapopan, Jalisco
  - Pfizer Investigational Site, Mexico City, Mexico City
- Russia (2):
  - Pfizer Investigational Site, Arkhangelskaya Obl, Primorsky Raion
  - Pfizer Investigational Site, Khot'kovo
- Spain (2):
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Madrid
- Pfizer Investigational Site, Taipei, Taiwan
- Pfizer Investigational Site, Caracas, Distrito Federal, Venezuela

REFERENCES:
- [Derived] Bowden CL, Vieta E, Ice KS, Schwartz JH, Wang PP, Versavel M. Ziprasidone plus a mood stabilizer in subjects with bipolar I disorder: a 6-month, randomized, placebo-controlled, double-blind trial. J Clin Psychiatry. 2010 Feb;71(2):130-7. doi: 10.4088/JCP.09m05482yel. Epub 2010 Jan 26. PMID 20122373
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281137&StudyName=Safety%20and%20Maintenance%20of%20Effect%20of%20Ziprasidone%20Plus%20a%20Mood%20Stabilizer%20in%20Bipolar%20I%20Disorder%20%28manic%20or%20mixed%29

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial intended to be outpatient trial. Patients hospitalized at the screening visit due to disease under study were to be stable enough for outpatient status within approximately 5 days.
Pre-assignment Details: Period 1:open label stabilization (ziprasidone plus lithium or valproic acid mood stabilizer). Period 2:subjects stabilized for 8 weeks randomized to blinded treatment (ziprasidone plus mood stabilizer or placebo plus mood stabilizer). 241 completed Period 1, 238 summarized in Period 2: 1 subject not randomized to Period 2, 2 excluded as per note.
Groups:
- Period 1 Open Label Ziprasidone: 40 - 80 milligram (mg) ziprasidone twice/day (BID) plus mood stabilizer. Dose adjusted on basis of toleration and efficacy.
- Ziprasidone: Double-blind, randomized ziprasidone at the dose level received during the last 4 weeks of Open Label Period.
- Placebo: Double-blind,randomized to placebo plus mood stabilizer. Subjects were tapered off ziprasidone onto placebo by decreasing 20 mg BID every 2 days during the first week of Period 2
Period: Period 1 Open Label Ziprasidone
Arm/Group | Period 1 Open Label Ziprasidone | Ziprasidone | Placebo
Started | 584 (1 subject inappropriately randomized into 2 different sites. Data from this subject was excluded.) | 0 | 0
Completed | 241 (Subject excluded as described above is counted as 2; enrolled in 2 sites (2 identification numbers)) | 0 | 0
Not Completed | 343 | 0 | 0
Not completed — Lack of Efficacy | 31 | 0 | 0
Not completed — Laboratory Abnormality | 3 | 0 | 0
Not completed — Adverse Event | 148 | 0 | 0
Not completed — Lost to Follow-up | 35 | 0 | 0
Not completed — Withdrawal by Subject | 76 | 0 | 0
Not completed — Miscellaneous | 50 | 0 | 0
Period: Period 2 Double Blind
Arm/Group | Period 1 Open Label Ziprasidone | Ziprasidone | Placebo
Started | 0 (1 subject in Period 1 did not want to be randomized into Period 2) | 127 | 111
Completed | 0 | 84 | 54
Not Completed | 0 | 43 | 57
Not completed — Lack of Efficacy | 0 | 9 | 22
Not completed — Laboratory Abnormality | 0 | 1 | 0
Not completed — Adverse Event | 0 | 11 | 15
Not completed — Lost to Follow-up | 0 | 3 | 6
Not completed — Withdrawal by Subject | 0 | 9 | 9
Not completed — miscellaneous | 0 | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ziprasidone | Placebo | Total
Number analyzed (Participants) | 127 | 111 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (12.3) | 38.0 (11.6) | 38.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 58 | 109
  Male | 76 | 53 | 129

OUTCOME MEASURES:

1. Primary Outcome: Time to Intervention for a Mood Episode During Double Blind Period
Description: Time to Intervention for Mood Episode (TIME) while on randomized drug after at least 8 weeks of symptom reduction on open-label ziprasidone plus mood stabilizer. Mood episode considered to have occurred and subject discontinued if one or more of the following: Investigator (INV) decides discontinuation is in best interest of subject; loss of effect and/or change to treatment regimen (INV judgment); subject hospitalized for disease under study; Mania Rating Scale (MRS) and/or Montgomery-Asberg Rating Scale (MADRS) rating is ≥18 for 2 consecutive visits scheduled no more than 10 days apart.
Time Frame: Period 2: 24 weeks or time of early termination
Population: Intent to Treat (ITT):Subjects took at least 1 dose double blind medication and had at least 1 post randomization observation. Double Blind Period followed at least 8 weeks open-label ziprasidone plus mood stabilizer; 25 out of 127 and 36 out of 111 subjects had an intervention for a mood episode.
Measure: Mean (Standard Error); unit: Days
Groups:
- Ziprasidone: Randomized to Double Blind Therapy with Ziprasidone plus mood stabilizer
- Placebo: Randomized to Double Blind Therapy with Placebo plus mood stabilizer
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 127 | 111
Days | 172.159 (5.646) [7 to 201] | 143.133 (7.532)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Equality of Survival Curves across the treatment groups; Test type: Superiority or Other; p = 0.0104, Log Rank; alpha = 0.05 level of significance

2. Secondary Outcome: Time to Discontinuation for Any Reason During Double Blind Period 2
Description: Key Secondary endpoint is time to discontinuation for any reason. Profile of patients remaining in the trial over time.
Time Frame: Period 2: 24 weeks or time of early termination
Population: Intent to Treat (ITT). Number of participants who discontinued was 43 and 57 for ziprasidone and placebo, respectively.
Measure: Mean (Standard Error); unit: days
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 43 | 57
days | 153.526 (6.454) | 123.313 (7.524)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; alpha = 0.05 level of significance; Test type: Superiority or Other; p = 0.0047, Log Rank; No adjustment made for multiple comparisons

3. Secondary Outcome: Modified Time to Intervention for a Mood Episode (TIME)
Description: Time to intervention for a mood episode or time to discontinuation for treatment related adverse events, or death due to drug, or death due to disease. Mood episode considered to have occurred and subject discontinued if one or more of the following: Investigator (INV) decides discontinuation is in best interest of subject; loss of effect and/or change to treatment regimen (INV judgment); subject hospitalized for disease under study; Mania Rating Scale (MRS) and/or Montgomery-Asberg Rating Scale (MADRS) rating is ≥18 for 2 consecutive visits scheduled no more than 10 days apart.
Time Frame: Period 2: Week 24 or time of early termination
Population: Intent to Treat (ITT). 29 out of 127 ziprasidone subjects and 38 out of 111 placebo subjects met the modified criteria for an intervention for a mood episode
Measure: Mean (Standard Error); unit: Days
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 127 | 111
Days | 168.145 (5.857) | 140.325 (7.627)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; alpha = 0.05 level of significance; Test type: Superiority or Other; p = 0.0205, Log Rank — No adjustment made for multiple comparisons

4. Secondary Outcome: Change From Baseline in Mania Rating Scale (MRS) by Visit During Double Blind Period
Description: Period 2 Baseline = last observation in Period 1 to the start of Period 2. MRS is 11-item scale to measure mania; derived from Schedule for Affective Disorders and Schizophrenia-Change Behavior (SADS-CB). Subscales: Manic Syndrome (elevated mood, less need for sleep, excessive energy and activity, grandiosity), Behavior and Ideation (irritability, motor hyperactivity, accelerated speech, racing thoughts, poor judgment), and Impaired Insight. Racing thoughts range=0 to 2 (highest level of abnormal=2); all other items 0 to 5 (highest level of abnormal=5). Higher score = greater abnormality.
Time Frame: Period 2: Weeks 1 - 24 or time of early termination
Population: Intent to Treat (ITT); (n) = number of subjects with analyzable data at observation for ziprasidone and placebo, respectively.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 127 | 111
scores on scale
  Week 1 (n=121, 106) | -0.2 (3.0) | 0.8 (5.1)
  Week 2 (n=116, 95) | -0.4 (4.2) | -0.1 (4.7)
  Week 4 (n=117,95) | -0.6 (3.7) | 0.2 (5.4)
  Week 8 (n=107, 79) | -0.3 (5.7) | 0.8 (5.4)
  Week 12 (n=98, 70) | -1.0 (4.3) | 1.2 (8.2)
  Week 16 (n=94,65) | -1.4 (4.3) | 1.2 (6.3)
  Week 20 (n=84, 58) | -1.1 (6.5) | 0.2 (5.1)
  Week 24 (n=85,53) | -1.1 (5.5) | 0.3 (4.2)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Week 1: Difference in Change during Period 2 MMRM ANCOVA: center, subject within center as random effects; treatment, visit, visit by treatment interaction as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.1247, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.85, Standard Error of Mean 0.55 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; Week 2 mixed effects repeated measures analysis of covariance (MMRM ANCOVA): center, subject within center as random effects; treatment, visit, visit by treatment interaction as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.7515, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.20, Standard Error of Mean 0.62 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; Week 4 mixed effects repeated measures analysis of covariance (MMRM ANCOVA): center, subject within center as random effects; treatment, visit, visit by treatment interaction as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.3074, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.63, Standard Error of Mean 0.62 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 4: Comparison: Ziprasidone vs Placebo; Week 8 mixed effects repeated measures analysis of covariance (MMRM ANCOVA): center, subject within center as random effects; treatment, visit, visit by treatment interaction as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.0758, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -1.25, Standard Error of Mean 0.71 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 5: Comparison: Ziprasidone vs Placebo; Week 12 mixed effects repeated measures analysis of covariance (MMRM ANCOVA): center, subject within center as random effects; treatment, visit, visit by treatment interaction as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.0162, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -1.98, Standard Error of Mean 0.82 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 6: Comparison: Ziprasidone vs Placebo; Week 16 mixed effects repeated measures analysis of covariance (MMRM ANCOVA): center, subject within center as random effects; treatment, visit, visit by treatment interaction as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.0003, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -3.01, Standard Error of Mean 0.83 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 7: Comparison: Ziprasidone vs Placebo; Week 20 mixed effects repeated measures analysis of covariance (MMRM ANCOVA): center, subject within center as random effects; treatment, visit, visit by treatment interaction as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.0242, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -2.21, Standard Error of Mean 0.98 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 8: Comparison: Ziprasidone vs Placebo; Week 24 mixed effects repeated measures analysis of covariance (MMRM ANCOVA): center, subject within center as random effects; treatment, visit, visit by treatment interaction as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.0161, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -1.71, Standard Error of Mean 0.71 — Mean Difference (Final Values) = Least Squares Mean

5. Secondary Outcome: Change From Baseline in Clinical Global Impression Severity (CGI-S) Score by Visit During Double Blind Period
Description: Baseline for Period 2 is the last observation in Period 1 to the start of Period 2. Clinical Global Impression Severity Score is 7-item scale rates severity of illness from 0=not assessed, 1= normal to 7=most extremely ill.
Time Frame: Period 2: Weeks 1 - 24 or time of early termination
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 127 | 111
scores on scale
  Week 1 (n=122, 106) | 0.1 (0.7) | 0.3 (1.0)
  Week 2 (n=117, 95) | 0.2 (0.9) | 0.2 (1.0)
  Week 4 (n=117, 95) | -0.0 (0.7) | 0.1 (0.9)
  Week 8 (n=107, 79) | -0.0 (0.8) | -0.1 (0.8)
  Week 12 (n=98, 70) | -0.1 (0.9) | 0.0 (1.1)
  Week 16 (n=94, 65) | -0.1 (0.9) | 0.0 (1.1)
  Week 20 (n=83, 58) | -0.1 (0.9) | -0.2 (1.0)
  Week 24 (n=85, 53) | -0.2 (1.0) | -0.2 (1.0)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Week 1 mixed effects repeated measures analysis of covariance (MMRM ANCOVA): center, subject within center as random effects; treatment, visit, visit by treatment interaction as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.0088, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.24, Standard Error of Mean 0.09 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.3677, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.11, Standard Error of Mean 0.13 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.0734, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.18, Standard Error of Mean 0.10 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 4: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.9166, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.01, Standard Error of Mean 0.11 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 5: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.2791, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.14, Standard Error of Mean 0.13 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 6: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.1460, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.23, Standard Error of Mean 0.16 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 7: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.7301, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.05, Standard Error of Mean 0.15 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 8: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p = 0.8162, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.03, Standard Error of Mean 0.14 — Mean Difference (Final Values) = Least Squares Mean

6. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Score by Visit During Double Blind Period
Description: Clinical Global Impression measures 7 items in Global assessment of improvement in patient's condition; 0=not assessed, 1= very much improved to 7= very much worse.
Time Frame: Period 2: Weeks 1 - 24 or time of early termination
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 127 | 111
scores on scale
  Week 1 (n=122, 106) | 2.3 (1.2) | 2.8 (1.6)
  Week 2 (n=117, 95) | 2.4 (1.4) | 2.6 (1.6)
  Week 4 (n=117, 95 | 2.3 (1.2) | 2.5 (1.5)
  Week 8 (n=107, 79) | 2.3 (1.4) | 2.2 (1.2)
  Week 12 (n=98, 70) | 2.2 (1.3) | 2.2 (1.4)
  Week 16 (n=94, 65) | 2.3 (1.4) | 2.5 (1.5)
  Week 20 (n=83, 58) | 2.1 (1.4) | 2.1 (1.4)
  Week 24 (n=85, 53) | 2.2 (1.3) | 2.2 (1.4)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0013, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.48, Standard Error of Mean 0.15 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.1167, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.27, Standard Error of Mean 0.17 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.0188, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.40, Standard Error of Mean 0.17 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 4: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.3413, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.15, Standard Error of Mean 0.16 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 5: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.2760, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.18, Standard Error of Mean 0.16 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 6: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.0085, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.51, Standard Error of Mean 0.19 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 7: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.1317, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.27, Standard Error of Mean 0.18 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 8: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p = 0.1666, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.25, Standard Error of Mean 0.18 — Mean Difference (Final Values) = Least Squares Mean

7. Secondary Outcome: Change From Baseline in Montgomery-Asberg Rating Scale (MADRS) Score by Visit During Double Blind Period
Description: Baseline for Period 2 is the last observation in Period 1 to the start of Period 2. MADRS is 10-item instrument measuring depression: scales from 0=Normal to 6 = most abnormal.
Time Frame: Period 2: Weeks 1 - 24 or time of early termination
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 127 | 111
scores on scale
  Week 1 (n=121, 106) | -0.2 (4.9) | 2.7 (7.3)
  Week 2 (n=117, 95) | 1.1 (7.4) | 2.7 (7.1)
  Week 4 (n=117, 95) | -0.3 (5.3) | 1.6 (6.0)
  Week 8 (n=107, 79) | 0.4 (5.9) | 0.4 (5.3)
  Week 12 (n=98, 70) | 1.1 (5.9) | 0.6 (5.4)
  Week 16 (n=94,65) | 1.2 (6.3) | 0.4 (3.9)
  Week 20 (n=84, 58) | 0.5 (5.6) | -0.2 (4.9)
  Week 24 (n=85, 53) | 0.4 (6.4) | 1.0 (6.5)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0023, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -2.29, Standard Error of Mean 0.75 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.1412, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -1.34, Standard Error of Mean 0.91 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.0861, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -1.49, Standard Error of Mean 0.87 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 4: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.5992, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.43, Standard Error of Mean 0.82 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 5: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.5873, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = 0.41, Standard Error of Mean 0.76 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 6: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.2116, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = 0.97, Standard Error of Mean 0.78 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 7: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.1847, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = 0.90, Standard Error of Mean 0.68 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 8: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p = 0.9972, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.00, Standard Error of Mean 0.82 — Mean Difference (Final Values) = Least Squares Mean

8. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score by Visit During Double Blind Period
Description: Baseline for Period 2 is the last observation in Period 1 to the start of Period 2. Positive and Negative Syndrome Scale Total Score is 30-item scale measuring severity of psychopathology (16 items), positive symptoms (7 items) and negative symptoms (7 items); scale from 1 (absent) to 7 (extreme)
Time Frame: Period 2: Weeks 4 - 24 or time of early termination
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 127 | 111
scores on scale
  Week 4 (n=123, 98) | 0.4 (8.7) | 1.5 (6.9)
  Week 8 (n=107, 79) | -0.1 (8.3) | -0.8 (6.0)
  Week 12 (n=98, 70) | -0.1 (6.5) | 0.3 (9.4)
  Week 16 (n=94, 65) | -0.0 (7.1) | 0.7 (8.7)
  Week 20 (n=84, 58) | -0.2 (7.4) | -1.0 (6.1)
  Week 24 (n=85, 53) | -0.6 (8.0) | -0.9 (7.4)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.5954, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.49, Standard Error of Mean 0.93 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.3414, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = 0.89, Standard Error of Mean 0.93 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.9745, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = 0.04, Standard Error of Mean 1.23 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 4: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.5627, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.85, Standard Error of Mean 1.47 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 5: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.7410, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = 0.36, Standard Error of Mean 1.10 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 6: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p = 0.9632, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.04, Standard Error of Mean 0.88 — Mean Difference (Final Values) = Least Squares Mean

9. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Postive Scale by Visit During Double Blind Period
Description: Baseline for Period 2 is the last observation in Period 1 to the start of Period 2. Positive Scale is 7-items derived from PANSS; 1 (absent), 2 (minimal) to 7 (extreme).
Time Frame: Period 2: Weeks 4 - 24 or time of early termination
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 127 | 111
scores on scale
  Week 4 (n=123, 98) | 0.0 (1.6) | 0.1 (1.4)
  Week 8 (n=107, 79) | -0.2 (2.0) | -0.2 (1.9)
  Week 12 (n=98, 70) | -0.3 (1.7) | 0.3 (3.3)
  Week 16 (n=94, 65) | -0.4 (1.8) | 0.0 (2.1)
  Week 20 (n=84, 58) | -0.2 (2.2) | -0.1 (2.1)
  Week 24 (n=85, 53) | -0.2 (2.2) | -0.1 (2.1)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.9538, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = 0.01, Standard Error of Mean 0.22 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.8541, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = 0.05, Standard Error of Mean 0.25 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.1084, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.52, Standard Error of Mean 0.32 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 4: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.0380, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.56, Standard Error of Mean 0.27 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 5: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.2649, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.39, Standard Error of Mean 0.35 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 6: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p = 0.2394, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = -0.32, Standard Error of Mean 0.27 — Mean Difference (Final Values) = Least Squares Mean

10. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Negative Scale by Visit During Double Blind Period
Description: Baseline for Period 2 is the last observation in Period 1 to the start of Period 2. Negative Scale is 7 items derived from PANSS; scale is 1 (absent) to 7 (extreme).
Time Frame: Period 2: Weeks 4 - 24 or time of early termination
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 127 | 111
scores on scale
  Week 4 (n=123, 98) | 0.2 (3.1) | 0.4 (2.2)
  Week 8 (n=107, 79) | 0.2 (3.2) | -0.1 (1.8)
  Week 12 (n=98, 70) | 0.1 (2.5) | 0.1 (2.1)
  Week 16 (n=94, 65) | 0.3 (3.1) | 0.4 (2.6)
  Week 20 (n=84, 58) | -0.0 (2.3) | -0.4 (1.8)
  Week 24 (n=85, 53) | -0.1 (2.6) | -0.1 (2.1)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.8117, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = 0.07, Standard Error of Mean 0.29 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.0443, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = 0.51, Standard Error of Mean 0.26 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.3039, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = 0.29, Standard Error of Mean 0.28 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 4: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.9953, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = 0.00, Standard Deviation 0.46 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 5: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.1653, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = 0.44, Standard Error of Mean 0.32 — Mean Difference (Final Values) = Least Squares Mean
Statistical Analysis 6: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p = 0.5771, MMRM ANCOVA; MMRM ANCOVA = mixed effects repeated measures analysis of covariance; Mean Difference (Final Values) = 0.18, Standard Error of Mean 0.32 — Mean Difference (Final Values) = Least Squares Mean

ADVERSE EVENTS:
Arm/Group | Period 1 Open Label Ziprasidone | Ziprasidone | Placebo
Serious Adverse Events (participants affected / at risk) | 15 | 3 | 2
Other Adverse Events (participants affected / at risk) | 362 | 22 | 24
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Period 1 Open Label Ziprasidone | Ziprasidone | Placebo
Influenza (Infections and infestations) | 1/584 | 0/127 | 0/112
Arrhythmia (Cardiac disorders) | 0/584 | 1/127 | 0/112
Dystonia (Nervous system disorders) | 1/584 | 0/127 | 0/112
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/584 | 0/127 | 0/112
Affect lability (Psychiatric disorders) | 1/584 | 0/127 | 0/112
Anxiety (Psychiatric disorders) | 1/584 | 0/127 | 0/112
Bipolar I disorder (Psychiatric disorders) | 1/584 | 0/127 | 0/112
Bipolar disorder (Psychiatric disorders) | 2/584 | 0/127 | 0/112
Depression (Psychiatric disorders) | 1/584 | 0/127 | 0/112
Depression suicidal (Psychiatric disorders) | 1/584 | 0/127 | 0/112
Mania (Psychiatric disorders) | 2/584 | 0/127 | 2/112
Psychiatric decompensation (Psychiatric disorders) | 1/584 | 0/127 | 0/112
Psychotic disorder (Psychiatric disorders) | 1/584 | 0/127 | 0/112
Suicidal ideation (Psychiatric disorders) | 2/584 | 2/127 | 0/112
Suicide attempt (Psychiatric disorders) | 1/584 | 0/127 | 0/112
Thrombophlebitis (Vascular disorders) | 1/584 | 0/127 | 0/112
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Period 1 Open Label Ziprasidone | Ziprasidone | Placebo
Nausea (Gastrointestinal disorders) | 42/584 | 0/127 | 0/112
Fatigue (General disorders) | 44/584 | 0/127 | 0/112
Upper respiratory tract infection (Infections and infestations) | 0/584 | 5/127 | 6/112
Akathisia (Nervous system disorders) | 47/584 | 0/127 | 0/112
Dizziness (Nervous system disorders) | 49/584 | 0/127 | 0/112
Headache (Nervous system disorders) | 32/584 | 0/127 | 0/112
Sedation (Nervous system disorders) | 134/584 | 0/127 | 0/112
Somnolence (Nervous system disorders) | 99/584 | 0/127 | 0/112
Tremor (Nervous system disorders) | 73/584 | 8/127 | 4/112
Insomnia (Psychiatric disorders) | 59/584 | 7/127 | 12/112
Mania (Psychiatric disorders) | 0/584 | 3/127 | 6/112

LIMITATIONS AND CAVEATS:
This is a maintenance of effect design using a survival analysis methodology. In such a design it may be difficult to interpret timepoint by timepoint treatment group comparisons in MRS, CGI-S, CGI-I, MADRS, and PANSS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.